CLINICAL TRIAL: NCT02283697
Title: Assessment of Effectiveness of Counseling by a Registered Dietician on Low Salt Diet in Patients With Hypertension: A Pragmatic Clinical Trial.
Brief Title: Dietary Counseling to Reduce Salt Intake in Patients With High Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20142641
Record Dates: First submitted 2014-11-02; First posted 2014-11-05 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Hypertension
Keywords: hypertension; high blood pressure; sodium; prevention; dietary sodium; salt
MeSH Terms: conditions — Hypertension | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary Counseling (Experimental): Apart from standard care, an additional one on one (family members allowed) one hour long counseling by certified dietician who will assess the patient's dietary habits, endorse and describe the Dietary Approach to Stop Hypertension (DASH) diet, and will establish four weekly half an hour follow ups by telephone to address compliance and any question raised by patient and family members.
  Interventions: Behavioral: Dietary Counseling
- Control: Standard Care (Other): A standard endorsement of low salt diet and other non-pharmacological interventions such as moderation of alcohol intake, optimal body weight, daily exercise by hypertension nurse and physician
  Interventions: Other: Control: Standard Care

INTERVENTIONS:
Behavioral: Dietary Counseling — a standard endorsement of low salt diet and other non-pharmacological interventions such as moderation of alcohol intake, optimal body weight, daily exercise by hypertension nurse and physician AND an additional one on one (family members allowed) one hour long counseling by certified dietician who will assess the patient's dietary habits, endorse and describe the Dietary Approach to Stop Hypertension (DASH) diet, and will establish four weekly half an hour follow ups by telephone to address compliance and any question raised by patient and family members.
  Arms: Dietary Counseling
Other: Control: Standard Care — a standard endorsement of low salt diet and other non-pharmacological interventions such as moderation of alcohol intake, optimal body weight, daily exercise by hypertension nurse and physician
  Arms: Control: Standard Care

SUMMARY:
High salt diet increases risk of development of hypertension. In hypertensive patients, low salt diet decreases blood pressure. Not surprisingly public health authorities endorse low salt diet in hypertensive patients. But, surprisingly, average salt intake among adults in Canada remains stubbornly high. Low effectiveness of "fast counselling" by physicians and nurses on dietary salt is partly the culprit. Methods used in successful clinical trials (eg. provision of meals, community cooking sessions, many hours of counselling by dieticians) cannot be used in routine clinical practice. Hence the investigators propose a study on a pragmatic dietary counselling method suitable for clinical practice.

Hypertensive patients will be randomized to receive standard care (which includes counselling by the usual healthcare team, including doctors and nurses) or to receive additional counselling from a registered dietician. This counselling will include two components: a one hour counselling session, and 4, once-weekly telephone calls.

Effectiveness of this counselling will be measured by checking sodium in the urine from a 24 hour collection (which is a measure of dietary salt intake) at baseline and at 4 weeks. In addition, the investigators will also measure urinary sodium at 1 year, to assess if this effect of counselling persists over a longer time.

DETAILED DESCRIPTION:
The study is a pragmatic clinical trial, to test if additional counseling provided by a dietician results in a reduction in dietary sodium intake as compared to usual care.

The hypothesis is that additional individualized and focused counseling provided by a dietician will result in true change in dietary habits which will result in reduction of dietary salt intake at 4 weeks. Usual care has been shown in the past to be ineffective in actual reduction in dietary salt intake.

In the current model of treatment of hypertension, no funding is available for this additional counseling. Also, usual care has been shown to be ineffective in reducing salt intake. If positive, this study will help make the case for provision of dietary counseling, which can be made to funding bodies.

This will be a prospective, open-label with blinded endpoints, randomized controlled trial.

The intervention: One focused dietary counseling session, one hour long, with a registered dietician. In addition, this will be followed by four, once-weekly phone calls to provide reinforcement, and provide advice and support. This will be additional to usual care.

The control group will receive usual care, which is advice provided during their clinic visit by the hypertension specialists clinic registered nurses and hypertension specialist physicians.

Both groups will have additional measurements as follows:

* Baseline, 4 week and 12 month measurement of 24 hour urinary sodium and potassium
* Baseline, 4 week and 12 month measurement of 24 hour ambulatory blood pressure monitoring

The randomization process will consist of a computer generated random listing of the treatment allocations in variable permuted blocks of 4 and 6 with concealment of allocation. Though blinding of the patients is not possible for a behavioral intervention such as this, the assessment of the outcome, which is an objective measurement, will be done in a blinded fashion. All the study personnel collating and analyzing this data will be blinded to the treatment assignment. In addition, the lab personnel who will be measuring the urinary sodium (which is the primary outcome) will be blinded to treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 years) with hypertension defined as

* daytime BP readings above 140/90 mmHg (as assessed from 24-hr ABPM)) without treatment and/or
* any patient with treated hypertension irrespective of BP load based on 24-hr ABPM.

Exclusion Criteria:

* Pregnant patients and
* patients with following conditions:
* glomerular filtration rate <45 ml/min/1.75 m2,
* active infection,
* acute coronary syndrome,
* severe liver disease;
* psychiatric disorders and/or otherwise unable to sign consent;
* patients with clinically manifested generalized and/or cardiac volume overload who may require immediate changes in diuretic therapy (at the discretion of treating hypertension specialist).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Change in 24 hour urinary sodium excretion | 4 weeks
  Change in 24-hour urine sodium at 4 weeks
Change in 24 hour urinary sodium excretion | 12 months
  Change in 24-hour urine sodium at 12 months

SECONDARY OUTCOMES:
Change in 24 hour ambulatory blood pressure | 4 weeks and 12 months
  Changes in daytime average systolic BP by 24-hr Ambulatory Blood Pressure Machine
Change in 24 hour urinary potassium | 4 weeks and 12 months
  Changes in dietary potassium intake assessed from 24-hour urinary potassium
Change in body weight | 4 weeks and 12 months
  Change in body weight

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Ruzicka, MD PhD, Principal Investigator — Ottawa Hospital research Insititute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Ruzicka M, Ramsay T, Bugeja A, Edwards C, Fodor G, Kirby A, Magner P, McCormick B, van der Hoef G, Wagner J, Hiremath S. Does pragmatically structured outpatient dietary counselling reduce sodium intake in hypertensive patients? Study protocol for a randomized controlled trial. Trials. 2015 Jun 17;16:273. doi: 10.1186/s13063-015-0794-y. PMID 26081765